CLINICAL TRIAL: NCT01924494
Title: Gastrointestinal Tele-Endoscopy Project: Synchronous Tele-Endoscopy - A Clinical Feasibility Study of Implementation of EndoAlpha Platform in Gastrointestinal Endoscopy.
Brief Title: Gastro Intestinal Tele Endoscopy Project
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Soren Meisner, Consultant, Head of GI Endoscopy Unit, Bispebjerg Hospital
Other Study IDs: GITEP
Record Dates: First submitted 2012-08-16; First posted 2013-08-16 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Investigate the Potential Network Limitations; Validate the Technology for Later Clinical Use; Evaluate System Integration of EndoAlpha
Keywords: telemedicine, tele-endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Endoscopy procedures: Patients undergoing elective flexible gastrointestinal endoscopy procedures

SUMMARY:
Synchronous Tele-Endoscopy: A clinical feasibility study of gastrointestinal tele-endoscopy by implementing and evaluating synchronous tele-endoscopy using ENDOALPHA in a hospital based endoscopy unit. EndoAlpha will be used on the hospitals existing Intranet/LAN and the possibilities of tele-endoscopy on WAN through existing network, on separate dedicated line or through new established transmission lines, will be evaluated. The EndoAlpha system will be integrated in a highly advanced endoscopy procedure room. The system will integrate through LAN with doctor office, clinic conference and lecture room and GI pathologist room. Through either LAN or WAN, connection will be establish to a referral GI center in Denmark. Through WAN, connection will be established to doctor home and to an expert Spanish center.

DETAILED DESCRIPTION:
Evaluate the potential network (LAN +WAN) limitations for video transmission image quality and audio transmission (two-way) quality. Validate the tele-endoscopy technology for consulting and second opinion in diagnostic endoscopy and therapeutic endoscopy (teaching, training and supervision of basic and advanced therapeutic procedures).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective gastrointestinal endoscopic procedures

Exclusion Criteria:

* Age < 18 years or > 90 years
* Unwilling to participate (no informed consent)
* Not able to understand and read Danish
* Emergency endoscopic procedures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective gastrointestinal endoscopy procedures
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the potential network (LAN +WAN) limitations for video transmission image quality and audio transmission (two-way) quality. | 1 year

SECONDARY OUTCOMES:
Validate the tele-endoscopy technology for consulting and second opinion in diagnostic endoscopy and therapeutic endoscopy (teaching, training and supervision of basic and advanced therapeutic procedures). | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Bispebjerg Hospiatl, Copenhagen, Denmark